CLINICAL TRIAL: NCT05044364
Title: A Randomized, Single-blind, Positive Drug Parallel Controlled, Multi-center Clinical Study on the Efficacy and Safety of Clevidipine Butyrate Injection in the Treatment of Hypertensive Emergency and Sub-emergency
Brief Title: Clinical Study of Clevidipine Butyrate Injection in the Treatment of Hypertensive Emergency and Sub-emergency
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cevidipine Butyrate Injection
Record Dates: First submitted 2021-09-05; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Hypertensive Emergency
MeSH Terms: conditions — Hypertensive Crisis | interventions — Single-Blind Method

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- China clevidipine butyrate injection (Experimental): Yangtze River Pharmaceutical Group Co., Ltd.
  Interventions: Drug: This is a randomized, single-blind, parallel-controlled clinical study with the original research clevidipine butyrate injection as the positive control drug, which is an equivalence test.
- Original research clevidipine butyrate injection (Active Comparator): Fresenius Kabi Austria Gmb H (Austria)
  Interventions: Drug: This is a randomized, single-blind, parallel-controlled clinical study with the original research clevidipine butyrate injection as the positive control drug, which is an equivalence test.

INTERVENTIONS:
Drug: This is a randomized, single-blind, parallel-controlled clinical study with the original research clevidipine butyrate injection as the positive control drug, which is an equivalence test. — Patients with hypertensive emergency and hypertensive sub-emergency who are clinically diagnosed as unsuitable for oral antihypertensive treatment or oral antihypertensive treatment are ineffective, and require intravenous medication to quickly control their blood pressure. The qualified subjects will be randomly divided into groups according to the test protocol. The method of administration is to infuse clevidipine butyrate injection for emergency blood pressure reduction treatment to achieve rapid, effective and stable lowering of blood pressure to the target blood pressure, and prevent or reduce further damage to the target organ.

SUMMARY:
Emergency treatment warning of clevidipine butyrate butyrate injection or invalid medical treatment and verification of the effectiveness and safety of subacute.

DETAILED DESCRIPTION:
The goal of the research and research is 18 weeks ≤ years of age, age ≤ 75 years of age, males are not limited; thoughtful for patients who are not suitable for taking medications or treating oral medications and need to quickly control blood sugar in emergency and hypertension sub-emergency patients, who meet the following conditions One: ① Clinic systolic pressure (SBP)>180mmHg and/or clinic diastolic pressure (DBP)>120mmHg, with or without target organ damage; ②The degree of increase at the time of consultation did not reach SBP>180mmHg and or DBP> Patients with 180mmHg and or DBP>180mmHg but with indications of intravenous infusion of menstrual blood. According to the inflation method specified in the test protocol, clevidipine butyrate injection was infused for more urgent treatment to achieve rapid, effective, and slow reduction of blood sugar to the target blood sugar to prevent or start further organ damage.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ age ≤ 75 years old, men and women are not restricted;
2. Hypertensive emergency and hypertensive sub-emergency patients who are not suitable for oral antihypertensive treatment or oral antihypertensive treatment are ineffective and require intravenous medication to quickly control blood pressure, and meet one of the following conditions: ① Consultation systolic blood pressure (SBP)> Patients with 180mmHg and/or consulting room diastolic blood pressure (DBP)> 120mmHg, with or without target organ damage;

   ②Patients whose blood pressure is moderately elevated at the time of consultation, although SBP>180mmHg and/or DBP>120mmHg have not reached SBP>180mmHg and/or DBP>120mmHg, but the investigator has judged patients with indications for venous hypotension;
3. To participate in this clinical trial voluntarily, the subject (or legal representative) signs an informed consent form.

Exclusion Criteria:

1. Those who cannot receive intravenous infusion of antihypertensive drugs for 18 hours or more;
2. Patients with severe lipid metabolism abnormalities (such as triglycerides> 5mmol/L, familial hypercholesterolemia, lipid nephropathy, or acute pancreatitis accompanied by hyperlipidemia);
3. Patients who are known to have severe liver insufficiency or a history of liver failure or cirrhosis;
4. Patients who are known to be intolerant or allergic to study drugs or calcium channel blockers, or are allergic to the ingredients of study drug excipients, or are allergic to soybeans, soy products, eggs and egg products;
5. Patients with known or suspected severe aortic stenosis;
6. Those with a clear history of secondary hypertension (including: pheochromocytoma, primary aldosteronism, etc.);
7. Patients with known or suspected aortic dissection;
8. Those with a history of drug or alcohol abuse, and those with acute hypertension caused by drug overdose;
9. Pregnant or lactating women or patients who wish to have children during the trial period;
10. Patients who have participated in clinical trials of other drugs or devices in the past 30 days;
11. Patients who the investigator thinks are not suitable to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-10-11 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-10-10 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients whose systolic blood pressure dropped to the target range within 30 minutes of starting the infusion. | 30 minutes
  The percentage of patients whose systolic blood pressure dropped to the target range within 30 minutes of starting the infusion.

CONTACTS AND LOCATIONS:
Overall Officials: DONG SHAOHONG, 59, Principal Investigator — Shenzhen People's Hospital
Locations (2):
- China (2):
  - Shenzhen People' S Hospital, Shenzhen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No